CLINICAL TRIAL: NCT05949567
Title: Does Position Influence the Diagnosis of Detrusor Overactivity in a Neurological Population - a Concordance Study Between Lying and Sitting Position
Brief Title: Does Position Influence the Diagnosis of Detrusor Overactivity in a Neurological Population
Acronym: Cysto-position
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: APHP230769
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Urodynamic Exam; Neurologic Disorder
Keywords: Urodynamic exam; detrusor overactivity; positon
MeSH Terms: conditions — Nervous System Diseases; Urinary Bladder, Overactive | interventions — Sitting Position

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lying position first - then sitting position (Experimental)
  Interventions: Other: urodynamic exam in sitting and lying position
- Sitting position first - then lying position (Experimental)
  Interventions: Other: urodynamic exam in sitting and lying position

INTERVENTIONS:
Other: urodynamic exam in sitting and lying position — Urodynamic exam with 1st filling in sitting or lying position. Then , during the same procedure, a second filling in the opposite position of the 1st filling (lying or sitting)

SUMMARY:
ICS (International Continence Society) recommendations published in 2017 recommend performing urodynamic examinations in the sitting or standing position. These recommendations are based on a review of the literature published in 2008, which has several limitations: heterogeneous populations, old and non-harmonized techniques, and very few neurological patients. It seems appropriate to focus on neurological patients and to examine the influence of position on the detection of detrusor overactivity in these patients.

The point here is to reexamine the ICS recommendations, which are not designed for neurological patients. Indeed, many patients suffering from Multiple Sclerosis (MS) or Parkinson's disease are unable to sit or stand for the duration of the urodynamic examination. The investigators would like to assess whether exploring sphincter disorders in the supine position is still interpretable.

This would enable us to define ICS good practice recommendations for a neurological population.

DETAILED DESCRIPTION:
1st consultation (selection - D-15):

* Targeted questioning of disorders, completion of USP self-questionnaire, and UPDRS or EDSS scales as part of care.
* Verification of ultrasound results (for men).
* Schedule Urodynamic Assessment as part of treatment.
* Verification of eligibility criteria
* Partial information of the patient (or relative/guardian/guardian if applicable) to limit bias, and a period of reflection prior to the urodynamic test to collect consent.

On the day of the Urodynamic Assessment (D0):

* Written, free and informed consent.
* Data collection by a physician trained in the study,
* Randomization of patient to determine starting position (lying or sitting) for urodynamic assessment (via CleanWeb).
* Urodynamic assessment according to ICS recommendations, with constant filling speed over the 2 fillings (50 ml/min), water filling - Laborie machine - T-Doc system in both positions in the order defined by randomization, and printout of curves.
* Entry of socio-demographic data.
* Curves reread by a doctor who had not performed the examination and who did not know the patient or the starting position (single blind).
* Completion of the paper file by the physician reading the curves, with the following data for position 1 and position 2:
* Volume at B1 and B3 (in ml)
* Basal bladder pressure (cm / H2O)
* Occurrence of CNID or mictional reflex arc (diagnosis of detrusor overactivity)
* Volume of leakage or 1st NIDC (Uninhibited Detrusor Contraction) (ml) or
* Bladder pressure at leakage (cm / H2O)
* Maximum bladder pressure (cm / H2O)
* Paper data entry on Excel database by a trained investigator declared on the study

ELIGIBILITY:
Inclusion Criteria:

* Patient with MS or neurologically confirmed Parkinson's disease, with indication for urodynamic assessment - 1st assessment
* Clinical overactive bladder syndrome with USP overactive bladder sub-score > or = 4 - Age ≥18 years
* In men: no prostatic hypertrophy on ultrasonography
* In women: no stress urinary incontinence (SUI); USP SUI subscore ≤ 2
* Affiliated with a social security scheme (excluding AME).
* Free and informed written consent

Exclusion Criteria:

* Opposition to the performance of a Urodynamic exam as part of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
concordance diagnosis of detrusor overactivity between lying and sitting position | 24 months
  Measurement concordance of detrusor pressures using the intraclass correlation coefficient statistic

SECONDARY OUTCOMES:
position influence on the overactive detrusor gravity between the 2 positions | 24 months
  Measurement of the concordance of detrusor overactivity diagnostic gravities during urodynamic assessments, between those performed in the supine position and those performed in the seated position. Concordance will be assessed using Cohen's Kappa statistic.
Evaluation of the diagnosis quality of the detrusor overactivity between the 2 position | 24 months
  Measurement of the diagnostic quality of urodynamic testing performed in the supine position in neurological patients to detect detrusor activity, with the seated position being the gold standard: estimation of sensitivity and specificity.
comparison of the distribution of detrusor overactivity diagnoses according to position. | 24 months
  Measurement of the association between position during urodynamic assessment and diagnosis of detrusor overactivity: comparison of the distribution of diagnoses of detrusor overactivity according to position.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical and Rehabilitation Medicine Pitié Salpêtrière Hospital, Paris, France, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, National Commission for Computing and Liberties) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.